CLINICAL TRIAL: NCT01469026
Title: The Value of Early PET/CT in Patients With Metastasising Cancer of Unknown Primary
Brief Title: CUP Project PET/CT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Krogh Rask, Medical doctor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: K36
Record Dates: First submitted 2011-10-28; First posted 2011-11-10 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Metastasising Cancer of Unknown Primary
MeSH Terms: interventions — Radiation; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early PET/CT (Active Comparator)
  Interventions: Radiation: PET/CT or Conventional diagnostics including CT
- Conventional diagnostics including CT (Active Comparator)
  Interventions: Radiation: PET/CT or Conventional diagnostics including CT

INTERVENTIONS:
Radiation: PET/CT or Conventional diagnostics including CT — Radiation:
  PET/CT. 4 MBq/kg (max. 400 MBq) 18F-flour-deoxyglucosegiven iv. 60 min. before PET/CT scan.
  CT. iv.contrast medium (Ultravist 370 mg I/ml).
  Other Names: Radiation:; Positron emission tomography; Computed tomography

SUMMARY:
The purpose is to elucidate the value of PET/CT applied early in the work-up of patients with a metastasising cancer of an unknown primary tumor.

The management of patients with metastasising cancer of unknown primary often includes various and a large number of radiographic studies and invasive procedures, but the occult primary tumor is detected in less than 20%.

Early PET/CT may be useful in Cancer of Unknown Primary (CUP) before expensive and invasive diagnostic procedures are carried out. The outcome may be higher tumor detection rate and quicker diagnosis, avoiding unnecessary, extensive procedures. Furthermore, a large number of the patients will receive treatment aimed at the correct diagnosis. Therefore, a prospective cost-effectiveness analysis is warranted.

DETAILED DESCRIPTION:
Background:

Every year, 800-1000 patients in Denmark are classified with a diagnosis of metastasising cancer of unknown primary (CUP). This corresponds to approximately 3 % percent of all new cancer cases on a national scale. The number is probably higher, since this is a heterogeneous group of patients that is not registered consistently. The prognosis is poor; the average survival is only approximately one year.

CUP is characterized by the finding of a metastasis the starting point of which (the primary tumour) is unknown. Typically, one finds an enlarged lymph node in the neck, a swelling in the throat or in the stomach, a filling in the skin or a tumour detected somewhere in the body during an X-Ray examination, an endoscopy or the like. In spite of a search applying multiple techniques, the primary tumour remains unknown in 70-80% of the patients.

A great number of patients experience a long and discontinuous examination sequence marked by various contacts with doctors, many examinations dispersed over many days and locations, as well as a lot of time wasted, because there exists no single option or institution that takes care of the patient and handles diagnostic procedures and treatment efficiently.

Treatment is often initiated too late, typically as a combination of several chemotherapeutics in order to cover different types of cancer simultaneously, but modern chemotherapeutical regimes have not increased the survival rate. The bad prognosis is undoubtedly due to the fact that the patients are diagnosed in an advanced phase. Alternatively, the primary tumour is not detected at all. This, in part, is due to the absence of any single agency in possession of the competence and responsibility to implement the work-up without delay, and maybe because one does not offer examination by the modality (PET/CT) which is most likely to detect the presence of cancer, its starting point and dispersion in an early stage.

Methods:

Patients will be randomized 1:1 to the diagnostic arms 'conventional diagnostics incl. CT' or 'early PET/CT' at study entry. Before study start, a randomization list will be prepared according to which the assignment of patients to the treatment arms will be performed.

The early PET/CT examination will be performed at the Department of Nuclear Medicine at Odense University Hospital (OUH) using the tracer [18F]-fluorodeoxyglucose (FDG). Patients will be requested to appear in fasting state (minimum 6 hours) and will be administered intravenously FDG which is a radioactively labeled glucose-analog which enters cells by known glucose transport systems. The usage of FDG as cancer tracer is based on the increased metabolism and glucose demand of rapidly growing and proliferating cells. FDG remains within cells since it does not metabolize.

The patients will be scanned from the base of the scull to mid thigh by an integrated PET/CT scanner (GE Healthcare DiscoveryTM STE). A standardized CT protocol is used (Smart mA 30-400 mA with a noise index of 18.0 and rotation time of 0.8 s., kV 120, reconstruction thickness of 3.75 mm), followed by a PET examination (recording time is 2.5 min pr. field of view). CT scanning will be done with intravenous contrast medium (Ultravist 370 mg I/ml). The effective dose will be 18-20 mSv from CT and 5-6 mSv from FDG PET. Every patient at the Department of Nuclear Medicine has their height and weight measured before PET/CT and the PET/CT examination must be started in the interval 60 ± 5 min. after injection of FDG. Serum glucose concentration is measured before injection of FDG and must not exceed 8 mmol/L (150 mg/dL) The first 40 patients with a negative FDG-PET/CT will have an extra, late scan (without new contrast and with the same FDG-injection). One half (20 patients) will be scanned after 3 hours and the second half (20 patients) will be scanned 4 hours after the injection of FDG. This is to examine whether there is late focal uptake in some patients due to slow and only slightly increased glucose uptake. If so, the standard time point of scanning will in the remaining patients be at 3 or 4 hours after the injection of FDG in order to optimize the chance of detecting also slow growing tumours and metastases.

Identification of the primary tumor:

The primary tumor will be confirmed by histopathological examination of relevant biopsy specimens.

Endpoints:

In order to evaluate the hypotheses, the following data will be collected for all patients retrospectively from the local patient report filing system FPAS:

1. Detection of primary tumor possible: yes/no (primary endpoint)
2. Time frame from inclusion into the study to detection of primary tumor.
3. Time frame from inclusion into the study to referral to palliative or curative treatment.
4. Time frame from inclusion into the study to end of follow-up or death.
5. Total score of Quality of Life instrument "SF-36".

Population:

All patients are recruited from the Emergency Department based on subjective selection at the discretion of a trained internal medicine specialist (KKP). The expected number of patients will be 220.

Ethics:

The risk of PET/CT consists in the extra radiation dose (5-6mSv, p 4), which the PET-examination adds to the patient beyond the dose from CT (18-20mSv). The dose of radiation from PET is insignificant (a total estimated risk: 1/10.000), while the estimated risk from the radiation dose of CT is 1/1000. The lifetime risk of developing cancer is 25%. Performing the PET/CT scan increases the lifetime risk from 25% to 25,1%.

The radiation dose which is used has never been proven to cause adverse effects. The increase in lifetime effect is considered acceptable when compared to the improvement in diagnostic yield, patient course and targeted treatment.

Patient information describing the study and providing sufficient information for patients to make an informed decision about their participation will be handed out to patients in written form.

The patients will have 24 hours to think it over before making the final decision whether or not to participate. Participation is voluntary and consent can at anytime be withdrawn without any consequences for the patient's future treatment.

The Informed Consent form will be signed by all participating patients and stored at the Department of Nuclear Medicine

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven cancer without identified origin at the time of examination.
2. Patients admitted to but not fitting into existing cancer package programs.
3. Patients with very serious, but unknown, disease, which might be cancer.

Exclusion Criteria:

1. Patient belongs to one of the existing cancer packages - state which one.
2. Suspected metastasis in the liver.
3. Suspected metastasis in the brain.
4. Prior PET/CT imaging showing multiple metastases with no identifiable primary.
5. Cancer treatment already started.
6. Estimated inability to collaborate - state reason.
7. Prior malignant disease.
8. Pregnancy.
9. The patient cannot read and understand Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
1. Detection of primary tumor possible: yes/no (primary endpoint) | Up to 24 hours
  The outcome is evaluated based on the project specified PET/CT compared to conventional diagnostic investigations including CT. - The evaluation of the PET/CT scan, primary tumor/non-primary tumor, is obtained by consensus of two nuclear medicine physicians with experience in PET/CT.

SECONDARY OUTCOMES:
2. Time frame from inclusion into the study to detection of primary tumor. | Up to 1 week
  The time frame is determined by the number of days from the date of inclusion to the date of description for the PET/CT or the date of description for conventional CT.
3. Time frame from inclusion into the study to referral to palliative or curative treatment. | Up to 4 weeks
  The time frame is determined by the number of days from the date of inclusion to the date of description for the PET/CT or the date of description for conventional CT.
4. Time frame from inclusion into the study to end of follow-up or death. | 36 months
  Patients are followed till death or 36 months post inclusion.
5. Total score of Quality of Life instrument "SF-36". | 36 months
  Quality of life evaluation is performed at 3-6-12 and 36 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Depatment of Nuclearmedicine, Odense, Denmark